CLINICAL TRIAL: NCT01205373
Title: A Phase I Trial to Investigate the Metabolism and Pharmacokinetics of an Open-label Single Dose of 400 mg [14C]BI 671800 HEA Administered as an Oral Solution of the Choline Salt in Healthy Male Volunteers.
Brief Title: A Phase I Trial to Investigate the Metabolism and Pharmacokinetics as Well as Safety and Tolerability of a Single Dose BI671800 HEA Administered as an Oral Solution of the Choline Salt in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1268.7; 2009-016370-32 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-09-17; First posted 2010-09-20 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
MeSH Terms: interventions — BI 671800

ARMS (1):
- BI 671800 high dose (Experimental): Oral drinking solution
  Interventions: Drug: BI 671800

INTERVENTIONS:
Drug: BI 671800 — High dose oral drinking solution

SUMMARY:
The main objectives of the present study are to investigate the basic pharmacokinetics of BI 671800, its major metabolite CD6384, and 14C-radioactivity, including mass balance, excretion pathways and metabolism following a single oral dose of 400 mg [14C]BI 671800 HEA to healthy male volunteers. Secondary objectives are to evaluate the safety and tolerability following a single oral dose of 400 mg [14C]BI 671800 HEA to healthy male volunteers.

ELIGIBILITY:
Inclusion criteria:

1. Healthy males according to a complete medical history, including the physical examination (to be performed at Day -1), vital signs (blood pressure, pulse rate), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
2. Age 18 to 55 years, inclusive
3. Body mass index 18.0 to 30.0 kg/m2, inclusive
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion criteria:

1. Any finding of the medical examination (including blood pressure, pulse rate, and ECG) deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
5. History of relevant orthostatic hypotension, fainting spells, or blackouts
6. Chronic or relevant acute infections
7. History of relevant allergy/hypersensitivity (including allergy to study drug or its excipients)
8. Use of any prescription drugs 30 days prior to screening.
9. Use of any over-the-counter, non-prescription preparations (including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations) within 7 days prior to Check-in, unless deemed acceptable by the Investigator
10. Participation in another trial with an investigational drug within 2 months prior to administration or during the trial
11. Smoker (>10 cigarettes or >3 cigars or >3 pipes/day) or positive urine cotinine test at screening and check-in (Day -1)
12. Inability to refrain from smoking during the stay in the trial centre
13. Alcohol abuse (more than on average 2 units of alcoholic beverages per day or more than 14 units per week. One unit equals 1 pint (285 mL) of beer or lager, 1 glass (125 mL) of wine, or one shot (25 mL) of 40% spirit, or positive urine alcohol test at screening or check-in (Day -1)
14. Drug abuse
15. Blood donation (>100 mL within 60 days prior to study drug administration or during the trial)
16. Excessive physical activity (within 1 week prior to administration or during the trial until follow-up examination)
17. Any laboratory value outside the reference range that is of clinical relevance according to the investigator
18. Inability to comply with dietary regimen of study centre
19. A marked baseline prolongation of QT or QTc interval, history of additional risk factors for torsade de pointes (e.g. heart failure, hypokalaemia, family history of long QT syndrome)
20. Veins unsuitable for blood sampling
21. Exposure to diagnostic radiation for occupational reasons or during participation in a clinical trial in the previous year (except dental X-rays and plain X-rays of thorax and bony skeleton [excluding spinal column])
22. Irregular defecation pattern (less than once per day)
23. Unwillingness to use adequate contraception (condom plus another form of contraception e.g. spermicide, oral contraceptive taken by female partner, sterilisation, intrauterine device) during the entire study from the time of the first intake of study drug until 3 months after the last intake
24. Any laboratory value outside the reference range that is of clinical relevance, especially repeated Alanine transaminase (ALT), Aspartate transaminase (AST), Gamma-glutamyltransferase (GGT), alkaline phosphatase, or total bilirubin above upper limit of normal at screening and not resolved before dosing
25. Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval within 10 days prior to administration or during the trial, and Cytochrome P-450 (CYP)2C8 substrates such as amiodarone, amodiaquine, paclitaxel, rosiglitazone, pioglitazone and repaglinide or CYP2C9 such as warfarin, tolbutamide, phenytoin, losartan, acenocoumarol within 1 month or six half lives (whichever is greater)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2010-09; Primary Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Individual time course profiles of 14C-radioactivity (in nmol eq/L or nmol eq/kg for faeces) in whole blood, plasma, urine, and faeces | up to 336 h post treatment
Individual time course profiles of BI 671800 and its major metabolite CD6384 in plasma and urine | up to 336 h post treatment
Rate and extent of excretion mass balance based on the total radioactivity in urine and faeces | up to 336 h post treatment
Elucidation of metabolite structures and identification of major metabolites in plasma, urine, and faeces (if feasible) in comparison with various animal species (to be presented in a separate report) | up to 336 h post treatment
Cblood cells/Cplasma ratio of 14C-radioactivity | up to 168 h post treatment
concentrations of BI 671800 and its metabolite CD6384 in plasma and urine | up to 336 h post treatment
concentrations of 14C-radioactivity in whole blood, plasma, urine, and faeces | up to 336 h post treatment

SECONDARY OUTCOMES:
Changes from Baseline in Vital signs (pulse rate) | up to 23 days post treatment
Changes from Baseline in Physical examination | up to 23 days post treatment
Changes from Baseline in Vital signs (blood pressure) | up to 23 days post treatment
Changes from Baseline in 12-lead electrocardiogram (ECG) | up to 23 days post treatment
Changes from Baseline in Clinical laboratory tests | up to 23 days post treatment
Occurrence of Adverse Events | up to 23 days post treatment
Assessment of tolerability by investigator | up to 23 days post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1268.7.001 Boehringer Ingelheim Investigational Site, Madison, Wisconsin, United States